CLINICAL TRIAL: NCT06401395
Title: Clinical Evaluation of A neW Management Strategy for Patients With pArKinson's disEase usiNg an Innovative telemonitorING Device : AWAKENING Study
Brief Title: Clinical Evaluation of A neW Management Strategy for Patients With pArKinson's disEase usiNg an Innovative telemonitorING (AWAKENING)
Acronym: AWAKENING
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: DIAMPARK (Industry)
Collaborators: Weprom (Other); Digital Medical Hub (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: DigiParkMonitor_1.0_Awakening; 2024-A00464-43 (Other: French Health Products Safety Agency)
Record Dates: First submitted 2024-05-02; First posted 2024-05-06 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-04

CONDITIONS: Parkinson Disease
Keywords: Parkinson disease; Telemonitoring; Symptom management; Quality of life
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control arm (No Intervention): conventional follow-up only, i.e. a consultation with the neurologist every 6 months
- Telemonitoring arm (Experimental): remote monitoring using the DIGIPARK MONITOR application in addition to conventional monitoring.
  Interventions: Device: DIGIPARK MONITOR

INTERVENTIONS:
Device: DIGIPARK MONITOR — remote monitoring application (containing a questionnaire to assess the patient's symptoms, adapted from the clinical examination using the MDS-UPDRS scale). This questionnaire will be completed weekly for 12 months via the DIGIPARK MONITOR application by the patient or caregiver.
  Arms: Telemonitoring arm

SUMMARY:
Parkinson's disease (PD) ranks second among neurodegenerative diseases and is a major cause of neurological motor disability. The number of PD cases doubled between 1990 and 2016. The consequences of PD, including an increased risk of falls, loss of autonomy and reduced quality of life, contribute to increased morbidity and mortality. The costs associated with falls in the elderly (a fortiori those with PD) and their consequences represent between 0.85% and 1.5% of total healthcare expenditure.

There is currently no cure for PD. Treatment is symptomatic and depends on the degree of functional impairment and the age of onset. After a period of stabilization (state phase) of varying length, the clinical situation worsens because of treatment-related motor complications (motor fluctuations, on/off phenomena, dyskinesias, under/overdosing) and the appearance or worsening of disease-specific signs linked to the pathogenic process. Treatment of motor complications involves constantly adjusting doses and dosing schedules to suit each individual case, and to take account of variations in the patient's motor status over the months. These adjustments must also take into account the non-motor signs of the disease, notably thymic fluctuations, treatment-related behavioral disorders, fatigue, sensory and pain disorders. Regular follow-up of patients is therefore essential to assess the evolution of their symptoms, adjust treatment, adapt therapeutic interventions and improve their quality of life. However, most consultations with the neurologist are bi-annual, and because of the long time lapse between two consultations, the practitioner often has only incomplete information on the evolution of symptoms.

To help fill these gaps, advances in digital health technologies, with the development of telemonitoring solutions, enable patients to be monitored remotely and provide a potentially more robust amount of information relating to the severity of the disease and its evolution over time. In this sense, remote monitoring in PD would enable the neurologist to readjust treatment at the right time and in the most appropriate way. This will be done by means of a weekly questionnaire (adapted from the clinical examination via the MDS-UPDRS scale) completed by the patient via a mobile application.

Remote monitoring of patients should improve their symptom management and quality of life, hence the interest in an intervention offering a remote monitoring service: DIGIPARK MONITOR.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years ;
* Parkinson's disease according to MDS diagnostic criteria ;
* Classified as stage 1.5 to 3 according to the Hoehn and Yahr stages ;
* Followed by a neurologist since at least one month;
* Equipped with a smartphone or a computer or tablet with internet/cellular data access via the latter (or with the caregiver) ;
* Resident on French territory affiliated to a social security scheme.

Exclusion Criteria:

* Person under guardianship, curatorship or safeguard of justice or any other administrative or judicial measure of deprivation of rights and freedom;
* Patient suffering from dementia, mental disorders, cognitive disorders, or psychiatric pathology that could compromise the patient's informed consent and/or compliance with the study protocol;
* Patient deemed non-autonomous by the investigator and without a caregiver;
* Patient already included in another interventional research study, with the exception of NS-PARK's "PRECISE-PD" cohort.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Clinical effectiveness of telemonitoring on symptom progression in PD patients assessed by Movement Disorder Society- Unified Parkinson's Disease Rating scale (MDS-UPDRS) | 6 months
  total clinical examination score using the Movement Disorder Society- Unified Parkinson's Disease Rating scale (MDS-UPDRS). Score range from 0 to 200. A high score indicates clinical deterioration

SECONDARY OUTCOMES:
Evolution of PD patients' symptoms assessed by Movement Disorder Society- Unified Parkinson's Disease Rating scale (MDS-UPDRS) | 12 months
  Total clinical examination score using the Movement Disorder Society- Unified Parkinson's Disease Rating scale (MDS-UPDRS). Score range from 0 to 200. A high score indicates clinical deterioration
Specific quality of Life assessed by Parkinson Disease Questionnaire (PD-Q39). | 12 months
  score of Parkinson Disease Questionnaire (PD-Q39). Score range from 0 to 100. A high score indicates a deterioration
General quality of Life assessed by EuroQol-5 dimensions questionnaire | 12 months
  Score of EuroQol-5 dimensions questionnaire. Score range from 0 to 100. A high score indicates a improvement
Organizational impact assessed by the number of consultation that led to a paramedical and/or drug treatment rehabilitation between semi-annual consultations | 12 months
  Percentage of patients who had a consultation that led to a paramedical and/or drug treatment rehabilitation between semi-annual consultations
Medico-economic impact | 12 months
  Average total cost at 12 months in each group
Usability assessed by System Usability Scale. | 12 months
  System Usability Scale. Score range from 1 to 100. A high score indicates a improvement
User's satisfaction assessed by a spécific questionnaire created for the study | 12 months
  Satisfaction questionnaire created specifically for the study.Score range from 1 to 100. A high score indicates a improvement

CONTACTS AND LOCATIONS:
Overall Officials: Adeline GIANINA, Principal Investigator — Medipole Hopital Mutualiste
Locations (10):
- France (10):
  - CHU Angers, Angers
  - CH Flayriat, Bourg-en-Bresse
  - CHU Caen, Caen
  - Clinique du Plateau, Clamart
  - CH Emile Roux, Le Puy-en-Velay
  - Clinique Beau Soleil, Montpellier
  - CHU Nice, Nice
  - CH de Troyes, Troyes
  - Hopital jean Bernard, Valenciennes
  - Médipole Hôpital Mutuliste, Villeurbanne

IPD SHARING:
Plan to Share IPD: No